CLINICAL TRIAL: NCT07401927
Title: The Effects of Preemptive Analgesic Protocols on Perioperative Pain Management in Laparoscopic Hysterectomy: A Prospective Observational Study
Brief Title: Preemptive Analgesia in Laparoscopic Hysterectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Dilek Yeniay, Anesthesiology and Reanimation physician, Giresun University
Other Study IDs: GOKAEK 2025/13/9
Record Dates: First submitted 2026-01-27; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Analgesia; Laparoscopic Hysterectomy
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group İ (İbuprofen): Patients who are administered ibuprofen pre-emptively analgesia, in accordance with routine clinical practice.
  Interventions: Drug: Ibuprofen
- Group P (Parasetamol): Patients who are administered parasetamol pre-emptively analgesia, in accordance with routine clinical practice.
  Interventions: Drug: Parasetamol

INTERVENTIONS:
Drug: Ibuprofen — Administered as part of standard institutional anesthesia practice.
  Other Names: ibuprofen 400 mg
  Groups: Group İ (İbuprofen)
Drug: Parasetamol — Administered as part of standard institutional anesthesia practice.
  Other Names: parasetamol 1 g
  Groups: Group P (Parasetamol)

SUMMARY:
The aim of this study is to evaluate the effects of ibuprofen and paracetamol administered for pre-emptive analgesia to patients undergoing laparoscopic hysterectomy on pain scores during the first 24 hours postoperatively, the amount of opioids consumed postoperatively, and adverse effects such as postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Patients who undergo laparoscopic hysterectomy surgery are administered certain treatment methods for postoperative analgesia. These applications are a routine part of the procedure. They are medically and ethically necessary. Postoperative analgesia applications are initiated during the intraoperative process and continued during the postoperative process. The analgesia protocol to be used is determined by the patient's characteristics and the anaesthetist's experience. Multimodal analgesia protocols are scientifically accepted methods. Preemptive analgesia, a method used for pain control that reduces the severity of pain caused by analgesics, delays the initial need for analgesia, and reduces the need for painkillers, is one of these protocols. This method, applied before surgical incision or tissue damage, covers a wide range, from first-line analgesics such as paracetamol and ibuprofen to opioids and peripheral and central blocks. The aim of this study is to evaluate the effects of ibuprofen and paracetamol administered for preemptive analgesia in patients undergoing laparoscopic hysterectomy on pain scores in the first 24 hours postoperatively, the amount of opioids consumed postoperatively, and adverse effects such as postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70
* ASA I-III patients
* Patients undergoing elective laparoscopic hysterectomy surgery

Exclusion Criteria:

* Emergency surgery
* Patients who require conversion to abdominal hysterectomy during the intraoperative period
* Those with severe liver or kidney failure, a history of long-term nonsteroidal anti-inflammatory and opioid analgesic use
* Those with a history of gastrointestinal bleeding, peptic ulcer or inflammatory bowel disease, diabetes or other neuropathic diseases
* Patients unable to use patient-controlled analgesia (PCA) devices

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients aged 18 to 70 who are scheduled to undergo laparoscopic hysterectomy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia | from the end of surgery up to 24 hours postopeartively
  Postoperative analgesia was assessed by measuring postoperative pain intensity using the Visual Analog Scale (VAS) and by recording cumulative opioid or rescue analgesic consumption.
  The Visual Analog Scale ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain.
  Lower pain scores and reduced analgesic requirements were considered indicators of better postoperative analgesia.

SECONDARY OUTCOMES:
İntraoperative analgesia | During surgery (from skin incision until the end of surgery)
  Intraoperative analgesia was assessed by evaluating hemodynamic responses to surgical stimuli, including changes in heart rate and mean arterial pressure, as well as the requirement for additional intraoperative analgesic agents.
  Stable hemodynamic parameters and a reduced need for supplemental analgesia were considered indicators of adequate intraoperative analgesia.stimuli, including changes in heart rate and mean arterial pressure, as well as the requirement for additional intraoperative analgesic agents. Stable hemodynamic parameters and reduced need for supplemental analgesia were considered indicators of adequate intraoperative analgesia.
Intraoperative hemodynamic instability | During surgery (from induction of anesthesia until the end of surgery)
  Intraoperative hemodynamic instability was assessed by continuous monitoring of heart rate and mean arterial pressure throughout the surgical procedure.
  Hemodynamic instability was defined as the occurrence of hypotension, hypertension, bradycardia, or tachycardia based on deviations from baseline values.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and confidentiality considerations